CLINICAL TRIAL: NCT05725525
Title: Feasibility of Internet Delivered Parent Child Interaction Therapy (AI I-PCIT) Real-Time Monitoring of Sleep and Behavior of Children 3-7 Years-Old Receiving Remote PCIT
Brief Title: A Study of Internet Delivered Parent Child Interaction Therapy
Acronym: AI I-PCIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Magdalena Romanowicz, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-009425
Record Dates: First submitted 2023-01-13; First posted 2023-02-13 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Disruptive Behavior
Keywords: Garmin Watch; Artificial Intelligence; PCIT; Telehealth; Technology; Decentralized Trial
MeSH Terms: conditions — Problem Behavior | interventions — Wearable Electronic Devices

STUDY DESIGN:
Masking Description: All participants will receive the same interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wearable Device Intervention (Other): An open label, non randomized trial that requires all participants to wear a Garmin watch throughout the course of the trial (~12 weeks).
  Interventions: Behavioral: Remote PCIT augmented with wearable devices

INTERVENTIONS:
Behavioral: Remote PCIT augmented with wearable devices — Participants will be enrolled in remote PCIT and be asked to wear a Garmin watch throughout the course of the study in order to measure biometric fluctuations

SUMMARY:
The purpose of this study is to learn more about how feasible remote parent child interaction therapy (PCIT) is for children with disruptive behaviors and how to augment treatment with wearable devices.

DETAILED DESCRIPTION:
Children with disruptive behaviors aged 3-7 will wear a Garmin watch throughout the course of the study (approximately 12 weeks). Artificial Intelligence (AI) will be applied to analyze the vitals provided by the watch to monitor for disruptive behavior. Parent and child will be enrolled in remote PCIT sessions throughout the course of the trial. This study will not require any in person visits, all materials will be mailed to the patients home or sent electronically. The study will analyze how the use of a wearable device throughout PCIT will help increase the benefit to both parent and child as measured by biometrics via Garmin and by questionnaires preformed throughout the trial.

ELIGIBILITY:
Inclusion Criteria - Children (Aged 3-7):

* Outpatients.
* Able to provide developmentally appropriate informed assent, and legal guardians able to provide informed consent.
* EBP Severity rated above the clinically significant range (≥120; T-score ≥ 60) (Eyberg Child Behavior Inventory- ECBI; Eyberg & Pincus, 1999).
* Families approached for participation will be asked to commit to complete the treatment:
* At least one primary caregiver and the identified child will have to be able to speak and understand English;
* Must have the ability, technology, and internet access for remote therapy/research visits.

Inclusion Criteria - Adults (Any age):

* Agree to wear Garmin watch.
* Able to provide informed consent.
* Able to speak and understand English.
* Has the ability, technology, and internet access for remote therapy/research visits.

Exclusion Criteria - Children:

* Formal diagnosis of Severe Intellectual disability, Autistic Spectrum Disorder Level 3, or a psychotic disorder for the child.
* Parents not consenting to the study.
* Parents or child is not able to adhere to the study protocol.
* A Child who is reasonable expected to be unable to tolerate wearing the Garmin device for at least 70% of the time during the day and night 70% of the days during the treatment (12 weeks). This is based on the principal investigator's discretion.
* Unable to speak and understand English.
* Refusal or withdrawal of consent, inability, or unwillingness to adhere to study procedures.
* Children in foster care.
* Does not have the ability, technology, and/or internet access for remote therapy/research visits.
* Need for more intensive behavioral treatments such as ER visit for behavioral dyscontrol or hospitalization will not be exclusionary or exit criteria.

Exclusion Criteria - Adults:

* Unable to speak and understand English.
* Refusal or withdrawal of consent, inability, or unwillingness to adhere to study procedures.

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
How wearing a Garmin watch will help the remote PCIT clinical outcomes | Through study completion, approximately 2 years
  Biometrics from the Garmin watch will be analyzed through Fitabase: step count, activity intensity, calories, heartrate, and respirations. This data will be compared throughout the study to see if factors trend down by the end of the trial. This would indicate that the child's behaviors were calmer at the end of the therapy when compared to the beginning.
Number of participants able to wear the Garmin watch throughout remote PCIT | Through study completion, approximately 2 years
  The study will measure how often participants are wearing the device by monitoring two platforms that are paired with the watch: Fitabase and Ilumivu. These platforms inform the study team with wear time of the watch by the participant. A measurement of at least 70% of the time will be deemed feasible/acceptable for young patient's ability to wear the watch during therapy.
Evaluating parental acceptance of remote PCIT augmented with a Garmin device | Through study completion, approximately 2 years
  At the end of therapy, the parent will receive an emailed survey asking about their opinions of the study technology and how it added to their child's therapy experience.

SECONDARY OUTCOMES:
Evaluating clinical improvement from remote PCIT in regards to sleep | Through study completion, approximately 2 years
  The study will collect parental rating scale measures of their child's sleep (PSQ). These reports will be collected weekly and will be compared throughout the course of therapy to see if parental reports of sleep gets better (length of time child is in bed and sleeping increases by the end of therapy).
Evaluating clinical improvement from remote PCIT in regards to parental reports of behavior accuracy of indirect behavioral measures from wearable devices to parental ratings | Through study completion, approximately 2 years
  The study will collect weekly parental ratings of their child's behavior (ECBI). These reports will be compared throughout the course of therapy to see if reports of the child's behavior is getting better throughout therapy.
Evaluating measured sleep data throughout remote PCIT | Through study completion, approximately 2 years
  The Garmin device will measure sleep cycle data (deep sleep, light sleep, REM sleep and hours awake). This data will be analyzed throughout participation to see if overall sleep time and quality increases with the amount of time spent in therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Romanowicz, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials